CLINICAL TRIAL: NCT00003162
Title: Randomized Trial of Palliative Radiation Therapy for Osseous Metastases: A Study of Palliation of Symptoms and Quality of Life
Brief Title: Radiation Therapy in Treating Patients With Bone Metastases From Breast or Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RTOG-9714; CDR0000065957; NCCTG-R9714; NCI-P97-0124
Record Dates: First submitted 1999-11-01; First posted 2003-04-18 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer; Metastatic Cancer; Pain; Prostate Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; stage IV prostate cancer; recurrent prostate cancer; bone metastases; pain
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Pain; Prostatic Neoplasms | interventions — Analgesia; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3.0 Gy x 10 fractions in two weeks (Active Comparator): 3.0 Gy x 10 fractions for a total dose of 30.0 Gy in two weeks
  Interventions: Procedure: pain therapy; Radiation: radiation therapy
- 8.0 Gy x 1 fraction (Experimental): 8.0 Gy x 1 fraction for a total dose of 8.0 Gy in a single dose
  Interventions: Procedure: pain therapy; Radiation: radiation therapy

INTERVENTIONS:
Procedure: pain therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which radiation therapy regimen is more effective for bone metastases.

PURPOSE: Randomized phase III trial to compare different radiation therapy regimens in treating patients who have bone metastases from breast or prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the ability of a single fraction of radiation therapy vs multiple fractions to provide complete pain relief in patients with painful bone metastases from breast or prostate cancer.
* Determine the frequency and duration of pain relief and narcotic relief after these treatments in these patient populations.
* Compare the effect on quality of life of these two treatments in these patient populations.
* Compare the incidence of pathologic fracture within the treatment fields after these two treatments in these patient populations.

OUTLINE: This is a randomized study.

Patients are assigned to 1 of 2 treatment arms. Arm I consists of radiation therapy delivered in 10 fractions over 2 weeks. Arm II consists of a single dose of radiation therapy. Any retreatment does not occur until at least 4 weeks after prior treatment unless there is an increase of 2 points on the pain score.

Patients are followed and quality of life is assessed at 2 and 4 weeks, then at 2, 3, 6, 9, and 12 months, every 6 months for the next 3 years, then annually until death.

PROJECTED ACCRUAL: This study will accrue 938 patients within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven breast or prostate cancer
* Radiographic evidence of bone metastasis within 8 weeks of study
* Eligible treatment sites:

  * Weight-bearing sites:

    * Pelvis (excluding pubis)
    * Femur
    * Sacrum and/or sacroiliac joints
    * Tibia
  * Non-weight-bearing sites:

    * Up to 5 consecutive cervical, thoracic, or lumbar vertebral bodies
    * Lumbosacral spine
    * Up to 3 consecutive ribs
    * Humerus
    * Fibula
    * Radius with/without ulna
    * Clavicle
    * Scapula
    * Pubis
  * If multiple sites are treated, site is included as weight bearing if any of the sites include the pelvis, sacrum, femur, or tibia
* Worst pain score of at least 5 on a scale of 10
* No skull, feet, or hand metastases
* No spinal cord or cauda equina compression/effacement in vertebral metastases
* Multiple sites eligible if they can be included in no greater than 3 treatment sites

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 40-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No impending fracture of the treatment site
* No hematologic primary malignancies
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No change in immunotherapy within 30 days

Chemotherapy:

* No change in chemotherapy within 30 days

Endocrine therapy:

* No change in hormonal therapy within 30 days

Radiotherapy:

* No prior radiation therapy to treatment area
* At least 30 days since systemic radiotherapy (Sr 89)

Surgery:

* No prior palliative surgery to treatment area
* No planned surgical fixation of the bone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 949 (Actual)
Dates: Start 1998-02; Primary Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William F. Hartsell, MD, Study Chair — Advocate Lutheran General Hospital; Ivy A. Petersen, MD, Study Chair — Mayo Clinic
Locations (253):
- United States (234):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscaloosa, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mount Diablo Medical Center, Concord, California
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Sutter Health West Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center, Pasadena, California
  - Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Inc., San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - St. Joseph's Regional Health System, Stockton, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Saint Mary's Hospital and Medical Center, Grand Junction, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Howard University Cancer Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center, Gainesville, Florida
  - Edna Williams Cancer Treatment Center, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Clarian Health Partners Inc., Indianapolis, Indiana
  - Regional Cancer Center, Indianapolis, Indiana
  - Oncology Institute of Greater Lafayette, Lafayette, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Lexington Clinic Cancer Center, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - Nebraska Health System, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Cooper Cancer Institute, Camden, New Jersey
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Kimball Medical Center, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Capital Health System at Mercer, Trenton, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Radiation Oncology Associates of Albuquerque, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Lourdes Regional Cancer Center, Binghamton, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Finger Lakes Radiation Oncology Center, Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - University of Rochester Cancer Center, Rochester, New York
  - North Shore Radiation Oncology, Setauket, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Medcenter One Health System, Bismarck, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Regional Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Cancer Center, East Stroudsburg, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Cancer Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon-Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - CCOP - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - All Saints Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (19):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Konski A, James J, Hartsell W, Leibenhaut MH, Janjan N, Curran W, Roach M, Watkins-Bruner D. Economic analysis of radiation therapy oncology group 97-14: multiple versus single fraction radiation treatment of patients with bone metastases. Am J Clin Oncol. 2009 Aug;32(4):423-8. doi: 10.1097/COC.0b013e31818da9f7. PMID 19546803
- [Background] Bruner DW. Outcomes research in cancer symptom management trials: the Radiation Therapy Oncology Group (RTOG) conceptual model. J Natl Cancer Inst Monogr. 2007;(37):12-5. doi: 10.1093/jncimonographs/lgm004. PMID 17951225
- [Background] Juliano JJ, Reddy CA, Videtic GMM: How fast does practice change? A single-institution experience in utilization of a single fraction for palliation of bone metastases before and after RTOG 9714. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-2561, S521-2, 2006.
- [Result] Chow E, James J, Barsevick A, Hartsell W, Ratcliffe S, Scarantino C, Ivker R, Roach M, Suh J, Petersen I, Konski A, Demas W, Bruner D. Functional interference clusters in cancer patients with bone metastases: a secondary analysis of RTOG 9714. Int J Radiat Oncol Biol Phys. 2010 Apr;76(5):1507-11. doi: 10.1016/j.ijrobp.2009.04.024. Epub 2009 Jul 23. PMID 19632065
- [Result] Howell DD, James JL, Hartsell WF, et al.: Randomized trial of short-course versus long-course radiotherapy for palliation of painful vertebral bone metastases: A retrospective analysis of RTOG 97-14. [Abstract] J Clin Oncol 27 (Suppl 15): A-9521, 2009.
- [Result] Hartsell WF, Desilvio M, Bruner DW, Scarantino C, Ivker R, Roach M 3rd, Suh J, Demas WF, Movsas B, Petersen IA, Konski AA. Can physicians accurately predict survival time in patients with metastatic cancer? Analysis of RTOG 97-14. J Palliat Med. 2008 Jun;11(5):723-8. doi: 10.1089/jpm.2007.0259. PMID 18588404
- [Result] Konski A, Desilvio M, Hartsell W, Watkins-Bruner D, Coyne J, Scarantino C, Janjan N. Continuing evidence for poorer treatment outcomes for single male patients: retreatment data from RTOG 97-14. Int J Radiat Oncol Biol Phys. 2006 Sep 1;66(1):229-33. doi: 10.1016/j.ijrobp.2006.04.005. Epub 2006 Jul 11. PMID 16814950
- [Result] Hartsell WF, Scott CB, Bruner DW, Scarantino CW, Ivker RA, Roach M 3rd, Suh JH, Demas WF, Movsas B, Petersen IA, Konski AA, Cleeland CS, Janjan NA, DeSilvio M. Randomized trial of short- versus long-course radiotherapy for palliation of painful bone metastases. J Natl Cancer Inst. 2005 Jun 1;97(11):798-804. doi: 10.1093/jnci/dji139. PMID 15928300
- [Result] Hartsell WF, Winter K, Bruner DW, et al.: Breast cancer patients have better outcomes than prostate cancer patients for palliation of painful bone metastases: results of RTOG 97-14. [Abstract] J Clin Oncol 23 (Suppl 16): A-6073, 546s, 2005.
- [Result] Bruner DW, Winter K, Hartsell W, et al.: Prospective health-related quality of life valuations (utilities) of 8 Gy in 1 fraction vs 30 Gy in 10 fractions for palliation of painful bone metastases: preliminary results of RTOG 97-14. [Abstract] Int J Radiat Oncol Biol Phys 60 (1 Suppl 1): A-23, S142, 2004.
- [Result] Hartsell WF, Scott C, Bruner DW, et al.: Phase III randomized trial of 8 Gy in 1 fraction vs. 30 Gy in 10 fractions for palliation of painful bone metastases: preliminary results of RTOG 97-14. [Abstract] Int J Radiat Oncol Biol Phys 57 (2 Suppl): S124, 2003.